CLINICAL TRIAL: NCT02554916
Title: Effectiveness of Rehabilitation Interventions for Mobility Impairment in Parkinson's Disease
Brief Title: Locomotor Adaptation Training to Prevent Mobility Disability
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400915-N; 1R21AG048133-01A1 (NIH)
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Age-related Mobility Decline
Keywords: Mobility decline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dual-belt Exercise: The participants assigned to this group will use the dual-belt treadmill 3 times a week for 16 weeks.
  Interventions: Behavioral: Dual-Belt Exercise; Device: Dual-Belt Treadmill
- Treadmill Exercise: The participants assigned to this group will use the treadmill 3 times a week for 16 weeks.
  Interventions: Behavioral: Treadmill Exercise; Device: Dual-Belt Treadmill
- Usual Care: The participants assigned to this group will not use the treadmills.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Dual-Belt Exercise — The dual-belted exercise treadmill can control the speeds of the right and left legs individually. When asymmetric, the dual-belt treadmill imposes mechanical and sensory perturbations independently to each leg such that the central nervous system (CNS) must solve and adapt to the challenge to maintain walking.
  Other Names: Dual-Belt Treadmill
  Groups: Dual-belt Exercise
Behavioral: Treadmill Exercise — The treadmill exercise will maintain the speed of the right and left leg together while walking.
  Groups: Treadmill Exercise
Other: Usual Care — This group will not be assigned to a treadmill but is as a non-exercising control group.
  Groups: Usual Care
Device: Dual-Belt Treadmill
  Groups: Dual-belt Exercise; Treadmill Exercise

SUMMARY:
This is an exploratory study designed to investigate the effects of aerobic dual belt treadmill walking versus traditional treadmill exercise on gait performance and functional capacity in older adults at risk for mobility disability. Identifying the relationship between aerobic treadmill exercise (dual belt or traditional) and the recovery of walking abilities will serve to optimize current rehabilitation approaches.

DETAILED DESCRIPTION:
Participants will be forty-eight older adults with pre-clinical mobility disability who will be randomized into one of three intervention groups: dual-belt treadmill exercise, traditional treadmill exercise, or non-contact control.

Prior to and following 16 weeks of therapy, we will observe the participants' performing several functional movements (walking, standing from sitting, sitting from standing, walking up and down stairs) and measure their muscular activity. These performance-based measures will be obtained to determine whether their movement function improves as a result of therapeutic intervention. The participants' absolute performance on any of these tasks does not matter as much as that they make the very best effort on each of the tests. They are welcome to take a break at any point in the testing or training.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Gait Speed of ≤ 1m/s
* Summary score 7-10 on the Short Physical Performance Battery, indicating mild to moderate impairment
* Sedentary as defined by reporting <20 min/wk of performing regular physical activity in the past month and <125 min/wk of moderate physical activity on the CHAMPS-18 questionnaire
* Willingness to be randomized to any of the treatment groups

Exclusion Criteria:

* Failure to provide informed consent
* Planned surgery in next year
* Hospitalization within the past 6 months
* Smoker > 1 pack per day
* Significant cognitive impairment, defined as a known diagnosis of dementia or a Modified Mini-Mental State score <24
* Significant cognitive executive impairment, defined as a Montreal Cognitive Assessment (MoCA) score of<25
* Progressive, degenerative neurologic disease, e.g., Parkinson's Disease, multiple sclerosis, Amyotrophic lateral sclerosis (ALS)
* Severe rheumatologic or orthopedic diseases, e.g., awaiting joint replacement, active inflammatory disease
* Terminal illness with life expectancy less than 12 mos, as determined by a physician
* Severe pulmonary disease, requiring either steroid pills or injections or the use of supplemental oxygen
* Severe cardiac disease, including New York Heart Association Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina;
* Other significant co-morbid disease that would impair ability to participate in the exercise-based intervention, e.g. renal failure on hemodialysis, severe psychiatric disorder (e.g. bipolar, schizophrenia), excessive alcohol use (>14 drinks per wk); persons with depression will not be excluded
* Develops chest pain or severe shortness of breath during exercise test
* Unable to communicate because of severe hearing loss or speech disorder or language barrier
* Lives outside of the study site or is planning to move out of the area in next year or leave the area for >1 month during the next year
* Severe diabetes, requiring use of insulin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults with sedentary lifestyle willing to be be randomized to and treatment groups.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2010-07; Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change in Gait Speed | baseline and up to 6 weeks following the intervention
  Gait speed will be determined from kinematic and kinetic measurement methods. A low value would indicate a slower walking speed compared to a higher value (faster walking speed).
Change in temporal variability | baseline and up to 6 weeks following the intervention
  Temporal will be determined from kinematic and kinetic measurement methods. Lower values correspond to better walking performance.
Change in spatial variability | baseline and up to 6 weeks following the intervention
  Spatial will be determined from kinematic and kinetic measurement methods. Lower values correspond to better walking performance.

SECONDARY OUTCOMES:
Change in physical performance | baseline and up to 6 weeks following the intervention
  Using the Short Physical Performance Battery. A score is generated from 0 (worst performance)-12 (best performance).
Change in cognitive impairment | baseline and up to 6 weeks following the intervention
  Using the Mini Mental State Exam. Each item has 5 possible points. Scores greater than or equal to 27 (out of 30) indicates normal cognition. Severe = <9, moderate = 10-18, and mild = 19-24 cognitive impairment.
Change in Cognitive impairment of executive function | baseline and up to 6 weeks following the intervention
  Using the Montreal Cognitive assessment. 30 items. A score of less than 26 on this assessment will indicate cognitive executive function.
Change in Disability | baseline and up to 6 weeks following the intervention
  The Pepper Assessment Tool for Disability will be used. Includes 5 subscales: mobility, transferring, upper extremity, instrumental and basic activities of daily living.
  Low scores indicate higher functioning and high independence. The Late-life function and Disability instrument will also be used. This has a 16-item disability component and a 32-item function component. Items are scored for 1-5 for function and 1-5 for frequency and extent of disability. Where high scores in frequency would represent more activity, and low scores in disability would represent less disabled.
Change in likelihood of falling | baseline and up to 6 weeks following the intervention
  Using the Dynamic Gait Index. This is an observational task that is scored on an ordinal scale. Total score per item is summed to a total score from 0(low level of function, high likelihood of falling)-24(high level of function, low likelihood of falling).
Change in knee extensor strength | baseline and up to 6 weeks following the intervention
  Using an isokinetic dynamometer, we will test Knee extensor strength. Peak torque will be calculated. A high value indicates more strength. Low values indicate less strength.
Change in ankle plantarflexor strength | baseline and up to 6 weeks following the intervention
  Using an isokinetic dynamometer, we will test ankle plantarflexor strength. Peak torque will be calculated. A high value indicates more strength. Low values indicate less strength.
Change in Timed up and Go | baseline and up to 6 weeks following the intervention
  Participants will be timed in seconds. More time to complete the task indicates low function, while less time indicates high function.
Change in timed chair rise | baseline and up to 6 weeks following the intervention
  Participants will be timed in seconds. More time to complete the task indicates low function, while less time indicates high function.
Change in timed stair climb | baseline and up to 6 weeks following the intervention
  Participants will be timed in seconds. More time to complete the task indicates low function, while less time indicates high function.
Change in energetic cost of walking | baseline and up to 6 weeks following the intervention
  This will be measured by: electrocardiogram, blood pressure, spirometry tests, and ratings of perceived exertion.
  The participant's maximal aerobic fitness, or oxygen consumption (VO2max) will be determined using a walking symptom-limited graded exercise test (GXT; modified walking incremental treadmill Naughton). All tests will follow the guidelines of the American College of Sports Medicine (ACSM) with electrocardiogram (ECG) heart monitoring and periodic blood pressure measures. Open-circuit spirometry will be used to determine VO2max and carbon dioxide production. Walking time until voluntary exhaustion or pain limitation will be recorded. Rating of perceived exertion (RPE) values will be collected at rest, at each exercise stage and during recovery. The treadmill tests will be performed at baseline and following the interventions.
Change in Ambulatory activity | baseline and up to 6 weeks following the intervention
  7 day assessment using an activity monitor. The device will count the number of steps taken.

CONTACTS AND LOCATIONS:
Overall Officials: Chris J Hass, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States